CLINICAL TRIAL: NCT07223177
Title: Philips FAST SpO2 Technology With Masimo Sensors for SpO2 Monitoring in the Neonatal, Infant, and Pediatric Populations
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Masimo Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: BERG0003
Record Dates: First submitted 2025-10-29; First posted 2025-10-31 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-01

CONDITIONS: SpO2

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Masimo Sensors (RD SET and/or LNCS) connected to Philips Monitors using Philips FAST SpO2 Algorithm (Experimental): All subjects are enrolled into this arm. All subjects will have blood oxygen measurements from:
  * non-invasive Masimo Sensors (RD SET and/or LNCS) connected to Philips Monitors using Philips FAST SpO2 Algorithm for blood oxygen measurements and
  * Masimo RD SET sensors connected to FDA-cleared pulse oximeter
  Interventions: Device: Masimo Sensor (RD SET and/or LNCS) connected to Philips Monitor using Philips FAST SpO2 Algorithm

INTERVENTIONS:
Device: Masimo Sensor (RD SET and/or LNCS) connected to Philips Monitor using Philips FAST SpO2 Algorithm — Subjects may use multiple Masimo sensors (RD SET and/or LNCS). All subjects will have at least one Masimo sensor (RD SET or LNCS) connected to Philips Monitors using Philips FAST SpO2 Algorithm

SUMMARY:
The objective of this study is to verify the form, fit and function of the Philips FAST technology with Masimo neonatal, infant and pediatric sensors for SpO2 monitoring in the respective indicated populations. The study design uses convenience sample data collection from neonatal, infant, and pediatric sensors within their respective indicated patient populations that have a range of different skin pigmentations, simultaneously with an FDA cleared pulse oximeter as a comparator.

ELIGIBILITY:
Inclusion Criteria:

* Subject falls within the indicated population for the Philips FAST SpO2 Monitor with the Masimo sensor.
* Subject is less than 22 years of age (pediatric subject per US FDA definition).

Exclusion Criteria:

* Subject has a skin condition or deformity at the planned sensor application site, which would preclude sensor placement and measurements as standard of care (e.g., psoriasis, eczema, angioma, scar tissue, burn, fungal infection, substantial skin breakdown).
* Confounders of pulse oximetry per sensor direction for use (DFU).
* Subject with distinct geographic variances in skin pigmentation (e.g., vitiligo), where the sensor is applied.
* Subject has an absence or deformities of limbs or severe edema, which would interfere with sensor application or prevent the proper fit of the sensors.
* Subject with nail polish or acrylic nails on the digits where sensor needs to be applied, who opts to not remove it.
* Subject with known allergic reactions to adhesive tapes.
* Subject is not suitable for the investigation at the discretion of the clinical research team.

Ages: 0 Years to 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-12-17 (Actual); Primary Completion 2026-06-05 (Estimated); Study Completion 2026-06-05 (Estimated)

PRIMARY OUTCOMES:
The acceptability of the quality of SpO2 signal obtained during non-invasive oxygen saturation monitoring using Philips FAST SpO2 technology with Masimo neonatal, infant, and pediatric sensors. Accuracy root mean square (ARMS) will be calculated. | 45 minutes

SECONDARY OUTCOMES:
The acceptability of the fit of sensor by visual observation of the emitter and detector alignment. | 45 minutes

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Paradigm Clinical Research, Modesto, California
  - Paradigm Clinical Research, San Diego, California